CLINICAL TRIAL: NCT03521245
Title: Molecular Pathway Activation Markers Predicting Efficacy of Trastuzumab Therapy for HER2-positive Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: OmicsWay Corp. (Industry)
Collaborators: Oncobox Ltd., Russia (Unknown); Vitamed LLC, Russia (Unknown); Republican Oncological Dispensary of Karelia Republic, Russia (Unknown)
Responsible Party: Principal Investigator, Anton A. Buzdin, Chief Scientific Officer, OmicsWay Corp.
Other Study IDs: OB0012018
Record Dates: First submitted 2018-04-28; First posted 2018-05-11 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: HER2-positive Breast Cancer
Keywords: breast cancer; epidermal growth factor receptor; HER2; EGFR; biomarkers; targeted therapy; NGS; RNAseq; mRNA; transcriptome analysis; signaling pathway; intracellular molecular pathway; Oncobox; trastuzumab
MeSH Terms: conditions — Breast Neoplasms | interventions — Sequence Analysis, RNA; RNA-Seq; Gene Expression Profiling; Trastuzumab; Drug Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Formalin-fixed, paraffin embedded pathological samples of breast cancer obtained during radical mastectomy or core needle biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Trastuzumab monotherapy: Her2-positive breast cancer patients treated with Trastuzumab (monotherapy)
  Interventions: Other: RNA sequencing; Other: Transcriptome analysis; Drug: Trastuzumab
- Chemotherapy plus Trastuzumab: Her2-positive breast cancer patients treated with Trastuzumab in combination with other regimens of chemotherapy
  Interventions: Other: RNA sequencing; Other: Transcriptome analysis; Drug: Trastuzumab; Drug: Chemotherapy

INTERVENTIONS:
Other: RNA sequencing — Next Generation Sequencing of RNA from tumor samples, rRNA-depleted.
  Other Names: RNA-seq
Other: Transcriptome analysis — Analysis of RNA-seq data using the Oncobox algorithm.
Drug: Trastuzumab — Standard Trastuzumab treatment regimen recommended for breast cancer
Drug: Chemotherapy — Standard chemotherapy regimen recommended for breast cancer
  Groups: Chemotherapy plus Trastuzumab

SUMMARY:
The purpose of the study is to identify molecular markers at the level of molecular pathway activation to predict efficacy of anti-HER2 therapy with Trastuzumab.

DETAILED DESCRIPTION:
Biopsy and/or surgical samples from Her2-positive breast cancer patients treated with Trastuzumab alone or in combinations with other regimens of chemotherapy with known clinical outcomes will be collected and subjected to mRNA sequencing. Expression profiles will be analysed using original bioinformatic platform Oncobox. Based on comparison of molecular pathways activation strength and clinical response to Trastuzumab and chemotherapy, this study aims to identify molecular markers predicting efficacy of therapy with Trastuzumab and the possibility of further relapse.

ELIGIBILITY:
Inclusion Criteria:

* adult females
* histologically confirmed HER2-positive breast cancer
* available FFPE samples of breast cancer tissue
* patients treated with Trastuzumab alone or in combination(s) with other regimens of chemotherapy with known outcome according to RECIST 1.1
* stage II or more
* patients who have signed an informed consent

Exclusion Criteria:

* less than 70% of intact tumor cells in available FFPE samples

Ages: 18 Years to 80 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Residents of North-Western and Central Parts of Russian Federation
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Tumor response by RECIST v1.1 or pathological response according to Chevallier system | 1 year
  Tumor response by RECIST v1.1 or pathological response according to Chevallier system

CONTACTS AND LOCATIONS:
Locations (4):
- OmicsWay Corp., Walnut, California, United States
- Russia (3):
  - Republican Oncological Dispensary of the Ministry of Healthcare of Karelia Republic, Petrozavodsk, Karelia Republic
  - Vitamed LLC, Moscow
  - "Oncobox" Ltd., Moscow

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol Statistical Analysis Plan (SAP) NGS data Clinical Study Report (CSR)
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months after trial completion, no end date
Access Criteria: Anyone